CLINICAL TRIAL: NCT03415178
Title: A Multicenter, Randomized, Open-label, Parallel-group Usability Study of the Commercial 1 mL Alirocumab Auto-injector Device (AI) and the New 2 mL Auto-injector Device (SYDNEY) in High or Very High Cardiovascular Risk Patients With Hypercholesterolemia Not Adequately Controlled With Their Lipid-Modifying Therapy
Brief Title: Usability Study of the Commercial Auto-injector Device and the New Auto-injector Device (SYDNEY) in Patients With High or Very High CV Risk With Hypercholesterolemia Not Adequately Controlled With Their Lipid-Modifying Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC14864; U1111-1186-3466 (Other: UTN)
Record Dates: First submitted 2018-01-04; First posted 2018-01-30 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Auto-Injector Device (AI) (Experimental): Alirocumab 300 milligram (mg) subcutaneous (SC) injection on Week 0 (Day 1), self-administered using AI device, on-site under supervision in the parallel arm treatment period of 4 weeks. From Week 4, participants switched to other arm of SYDNEY device to receive Alirocumab 300 mg, self- administered (unsupervised) using new auto-injector device (SYDNEY) every 4 weeks (Q4W) from Week 4 until Week 16 in the single arm treatment period added to lipid modifying therapy (LMT).
  Interventions: Drug: Alirocumab SAR236553; Device: Current auto-injector device (AI); Drug: Atorvastatin; Drug: Rosuvastatin
- New Auto-injector Device (SYDNEY) (Experimental): Alirocumab 300 mg SC injection on Week 0 (Day 1), self-administered using new auto-injector device (SYDNEY), on-site under supervision in the parallel arm treatment period of 4 weeks. From Week 4, same treatment (Alirocumab 300 mg) with the same device (SYDNEY) was self-administered, (unsupervised) Q4W until Week 16 in the single arm treatment period added to LMT. Duration of single arm treatment period was 12 weeks, i.e. from Week 4 to 16.
  Interventions: Drug: Alirocumab SAR236553; Device: New auto-injector device (SYDNEY); Drug: Atorvastatin; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Alirocumab SAR236553 — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous
Device: Current auto-injector device (AI) — Pharmaceutical form:
  Route of administration: Subcutaneous self-administration of alirocumab
  Arms: Auto-Injector Device (AI)
Device: New auto-injector device (SYDNEY) — Pharmaceutical form:
  Route of administration: Subcutaneous self-administration of alirocumab
  Arms: New Auto-injector Device (SYDNEY)
Drug: Atorvastatin — Pharmaceutical form:tablet Route of administration: oral
Drug: Rosuvastatin — Pharmaceutical form:tablet Route of administration: oral

SUMMARY:
Primary Objective:

To collect real-use (usability) data assessing the robustness and user interaction of the new alirocumab auto-injector device (which is referred to as SYDNEY), in unsupervised settings.

Secondary Objective:

Device-related:

* To collect real-use (usability) data assessing the robustness and user interaction of SYDNEY and the current alirocumab auto-injector device (which is referred to as AI) in supervised settings.

Pharmacokinetics:

* To compare alirocumab pharmacokinetics (PK) administered using SYDNEY and AI.
* To evaluate alirocumab PK administered using SYDNEY.

Anti-drug antibodies:

* To evaluate the development of anti-drug (alirocumab) antibodies (ADA).

Efficacy/pharmacodynamics:

* To compare the percent and absolute change in low-density lipoprotein cholesterol (LDL-C) using SYDNEY and AI.
* To evaluate the percent and absolute change in LDL-C using SYDNEY.

Safety:

* To evaluate the safety and tolerability of alirocumab using both SYDNEY and AI.

DETAILED DESCRIPTION:
Total study duration per participant was expected to be up to 18 weeks, with up to 2 weeks of screening period and 16 weeks of study treatment period.

ELIGIBILITY:
Inclusion criteria :

* Participants were in either category A or B (below), and were not adequately controlled with a stable daily dose of atorvastatin (20 mg or 40 mg), or rosuvastatin (10 mg or 20 mg) for at least 4 weeks prior to the screening visit (Week -2), with or without other LMT:

  * A. Participants with heterozygous familial hypercholesterolemia (heFH) (diagnosis based on either genotyping or clinical criteria) OR
  * B. Non-FH Participants at high or very high cardiovascular (CV) risk. High and very high cardiovascular risk participants included participants with coronary heart disease (CHD), non-CHD cardiovascular disease (CVD), and other risk factors.
* Participant willing and able to self-inject for the duration of the study.

Exclusion criteria:

* LDL-C <70 milligrams per deciliter (mg/dL) (<1.81 millimoles per litre [mmol/L]) at the screening visit.
* Currently taking a daily dose of statin that was not atorvastatin 20 mg or 40 mg, or rosuvastatin 10 mg or 20 mg.
* Not on a stable dose of LMT (including statin) for at least 4 weeks, prior to the screening visit and from screening to randomization.
* Having previously used any device for the proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor administration, or having participated in any clinical trial for a PCSK9 inhibitor.
* Fasting serum Triglyceride (TG) >400 mg/dL (>4.52 mmol/L) at the screening visit.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (13):
  - Investigational Site Number 8400024, Los Angeles, California
  - Investigational Site Number 8400007, Jacksonville, Florida
  - Investigational Site Number 8400017, Jacksonville, Florida
  - Investigational Site Number 8400013, Ponte Vedra, Florida
  - Investigational Site Number 8400014, Wellington, Florida
  - Investigational Site Number 8400001, West Des Moines, Iowa
  - Investigational Site Number 8400019, Topeka, Kansas
  - Investigational Site Number 8400006, Cincinnati, Ohio
  - Investigational Site Number 8400010, Cincinnati, Ohio
  - Investigational Site Number 8400022, Summerville, South Carolina
  - Investigational Site Number 8400026, Amarillo, Texas
  - Investigational Site Number 8400005, Richmond, Virginia
  - Investigational Site Number 8400027, Manitowoc, Wisconsin

REFERENCES:
- [Derived] Frias JP, Koren MJ, Loizeau V, Merino-Trigo A, Louie MJ, Raudenbush MA, Batsu I. The SYDNEY Device Study: A Multicenter, Randomized, Open-label Usability Study of a 2-mL Alirocumab Autoinjector Device. Clin Ther. 2020 Jan;42(1):94-107.e5. doi: 10.1016/j.clinthera.2019.11.008. Epub 2019 Dec 24. PMID 31879033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 13 centers in the United States. A total of 92 participants were screened on 29-March-2018 with randomization between 05 April 2018 and 12 April 18 of whom 23 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization to treatment arms was done centrally using treatment allocation system (Interactive Response Technology) in a 1:1 ratio (alirocumab from auto-injector device [AI] : alirocumab from new auto-injector device [SYDNEY]). A total of 69 participants were randomized.
Period: Parallel-Arm Period (up to Week 4)
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Started (Randomized) | 34 (Randomized) | 35 (Randomized)
Treated | 34 | 33
Completed | 34 (33 participants entered in single arm period & 1 participant decided not to enter single arm period.) | 33 (32 participants entered in single arm period & 1 participant decided not to enter single arm period.)
Not Completed | 0 | 2
Not completed — Randomized but not treated | 0 | 2
Period: Single Arm Period (up to Week 16)
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Started | 0 (Out of 34 participants from AI group, 33 participants entered entered in single arm period.) | 66 (65 (participants completed period 1) + 1 (randomized to SYDNEY arm but not treated in period 1).)
Completed | 0 | 65
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Auto-Injector Device (AI): Alirocumab 300 mg SC injection on Week 0 (Day 1), self-administered using AI device, on-site under supervision in the parallel arm treatment period of 4 weeks. From Week 4, participants switched to other arm of SYDNEY device to receive Alirocumab 300 mg, self- administered (unsupervised) using new auto-injector device (SYDNEY) Q4W from Week 4 until Week 16 in the single arm treatment period added to LMT.
- Total: Total of all reporting groups
Arm/Group | Auto-Injector Device (AI) | New Auto-injector Device (SYDNEY) | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.6) | 65.4 (8.1) | 65.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 15 | 26 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 24 | 31 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)] — Population: Calculated LDL-C in mg/dL from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/5]).
  Here, "Number analyzed" signifies number of participants with available data for this baseline measure.
  milligram per deciliter (mg/dL)
    number analyzed (Participants) | 34 | 34 | 68
    (all) | 98.6 (24.3) | 91.0 (15.0) | 94.8 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of SYDNEY-Associated Product Technical Complaints (PTCs) (Overall) at the Unsupervised Injections: Single-Arm Period
Description: SYDNEY-associated PTC was defined as any complaint reported on the participant complaint form that triggered an investigation by the device department and was categorized as either device-related, participant-related, or undetermined whether or not associated with an adverse event (AE). Overall category included total of all 3 types of PTCs. The percentage of SYDNEY-associated PTCs was calculated as: Number of PTCs / Number of unsupervised injections*100. The confidence interval (CI) was calculated using the Wilson score method.
Time Frame: From Week 4 up to Week 12
Population: Analysis was performed on safety population of the single-arm period which included all randomized participants who continued in the single-arm period and received at least 1 dose or part of a dose of investigational medicinal product (IMP) during this period.
Measure: Number (95% Confidence Interval); unit: percentage of PTCs
Units Other Than Participants: Number of unsupervised injections
Groups:
- New Auto-Injector Device (SYDNEY): All participants who were randomized to Alirocumab 300 mg SC injection using either AI device or SYDNEY in the parallel arm treatment period of 4 weeks and continued in single arm period, Alirocumab 300 mg self-administered (unsupervised) SC injection using SYDNEY device Q4W at Week 4, 8 and 12 in single arm period added to LMT. Duration of single arm treatment period was 12 weeks (i.e. from Week 4 to 16).
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 66
Number analyzed (Number of unsupervised injections) | 196
percentage of PTCs | 0.5 [0.0 to 3.2]

2. Primary Outcome: Percentage of SYDNEY-Associated Product Technical Complaints (PTCs) (by Type) at the Unsupervised Injections: Single-Arm Period
Description: SYDNEY-associated PTC was defined as any complaint reported on the participant complaint form that triggered an investigation by the device department and was categorized as either device-related, participant-related, or undetermined whether or not associated with an AE.
Time Frame: From Week 4 up to Week 12
Population: Analysis was performed on safety population of the single-arm period.
Measure: Number; unit: percentage of PTCs
Units Other Than Participants: Number of unsupervised injections
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 66
Number analyzed (Number of unsupervised injections) | 196
percentage of PTCs
  Device-related | 0
  Participant-related | 0.5
  Undetermined | 0

3. Secondary Outcome: Percentage of Participants With a SYDNEY or Current Auto-Injector (AI)-Associated Product Technical Complaint (PTCs) (Overall and by Type) at the Supervised Injections on Week 0 (Day 1): Parallel-Arm Period
Description: A PTC was defined as any complaint reported on the participant complaint form that triggered an investigation by the device department and was categorized as either device-related, participant-related, or undetermined, whether or not associated with an AE. Percentage of participants With a SYDNEY-associated PTC (for the reporting arm "Alirocumab from new auto-injector device") or Current AI-Associated PTCs (for the reporting arm "alirocumab from AI device") are reported.
Time Frame: Week 0 (Day 1)
Population: Analysis was performed on safety population of the parallel-arm period which included all randomized participants who received at least 1 dose or part of a dose of IMP during this period.
Measure: Number; unit: percentage of participants
Groups:
- Auto-Injector Device (AI): Alirocumab 300 mg SC injection on Week 0 (Day 1), self-administered using AI device, on-site under supervision in the parallel arm period of 4 weeks added to LMT.
- New Auto-Injector Device (SYDNEY): Alirocumab 300 mg SC injection on Week 0 (Day 1), self-administered using new auto-injector device (SYDNEY), on-site under supervision in the parallel arm period of 4 weeks added to LMT.
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 34 | 33
percentage of participants
  Overall | 0 | 0
  Type: Device-related | 0 | 0
  Type: Participant-related | 0 | 0
  Type: Undetermined | 0 | 0

4. Secondary Outcome: Percentage of Participants With SYDNEY-Associated Product Technical Complaint (PTCs) (Overall and by Type) at the Unsupervised Injections : Single-Arm Period
Description: A PTC was defined as any complaint reported on the participant complaint form that triggered an investigation by the device department and was categorized as either device-related, participant-related, or undetermined, whether or not associated with an AE. Percentage of Participants With a SYDNEY-associated PTC (for the reporting arm "Alirocumab from new auto-injector device [SYDNEY])" are reported.
Time Frame: From Week 4 up to Week 12
Population: Analysis was performed on safety population of the single-arm period.
Measure: Number; unit: percentage of participants
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 66
percentage of participants
  Overall | 1.5
  Type: Device-related | 0
  Type: Participant-related | 1.5
  Type: Undetermined | 0

5. Secondary Outcome: Injection Experience Questionnaire at Initial Supervised Injection: Overall Ease of Use Scores: Parallel-Arm Period
Description: Participants were given an injection experience questionnaire to complete after the self-injection they administered using SYDNEY device or current AI device on Day 1, for assessment of user experience and overall ease-of-use. The questionnaire included 9 questions about specific aspects of using the device. Overall ease of use was the 9th question, response of which ranged from 1 (very difficult) to 10 (very easy), with higher score indicated more ease of use.
Time Frame: Week 0 (Day 1)
Population: Analysis was performed on safety population of the parallel-arm period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auto-Injector Device (AI) | New Auto-injector Device (SYDNEY)
Number analyzed (Participants) | 34 | 33
score on a scale | 9.9 (0.2) | 9.8 (0.5)

6. Secondary Outcome: Patient Perspective Questionnaire After the Last Injection (at Week 12): Single-Arm Period
Description: The aim of the patient perspective questionnaire (completed by the participant after the last injection) was to generate data to support an understanding of the participant experience and satisfaction associated with use of the large volume SYDNEY to administer the 300 mg dose. The questionnaire consisted of 6 questions about level of satisfaction with various aspects of the SYDNEY; with response to each question ranging from 1 (very dissatisfied) to 10 (very satisfied), with higher scores indicated more satisfaction. An additional question (confidence that Sydney device was used correctly) regarding confidence of use of SYDNEY device in the study was evaluated on a scale of 10; where 1 being not at all confident, to 10 being very confident, higher scores indicated more confidence.
Time Frame: At Week 12
Population: Analysis was performed on safety population of the single-arm period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 66
score on a scale
  Size of the auto-injector | 9.7 (0.8)
  Ease of holding the auto-injector in hand | 9.8 (0.6)
  2-step operation:remove cap, press AI against skin | 9.9 (0.4)
  Length of time it took to complete the injection | 9.9 (0.3)
  Fact that needle is hidden prior & after injection | 10.0 (0.3)
  Once monthly injection | 10.0 (0.1)
  Confidence that Sydney device was used correctly | 9.9 (0.4)

7. Secondary Outcome: Injection-Treatment Acceptance Questionnaire (I-TAQ©) After Last Injection (at Week 12) - Overall Acceptance Scores: Single-Arm Period
Description: The I-TAQ© was a well-established and validated questionnaire to measure participant satisfaction with SC auto-injector devices. The I-TAQ© (completed by the participant after the last injection) was self-administered questionnaire administered to participants in order to measure their acceptance of the injection. The overall acceptance is one of the five domain scores. The overall acceptance score ranged from 0 to 100, with 0 indicating low acceptance and 100 indicating high acceptance.
Time Frame: At Week 12
Population: Analysis was performed on safety population of the single-arm period. Here, overall number of participants analyzed = participants who answered the I-TAQ.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 65
score on a scale | 93.08 (9.94)

8. Secondary Outcome: Maximum Serum Alirocumab Concentration Observed - Cmax : Parallel-Arm Period
Description: Cmax: Maximum serum concentration observed.
Time Frame: Pre-dose (Week 0) and on Day 7, 14 and 21
Population: Analysis was performed on pharmacokinetics (PK) population of the parallel-arm period which included all randomized participants who received at least 1 dose or part of a dose of IMP and had at least one evaluable blood sample for PK during this period. Here, "Overall number of participants analyzed" = participants evaluable for this PK measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 33 | 31
nanogram per milliliter (ng/mL) | 25800 (8430) | 26800 (8420)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alirocumab : Parallel-Arm Period
Description: Tmax: Time to reach Cmax.
Time Frame: Pre-dose (Week 0) and on Day 7, 14 and 21
Population: Analysis was performed on PK population of the parallel-arm period. Here, "Overall number of participants analyzed" = participants evaluable for this PK measure.
Measure: Median (Full Range); unit: days
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 33 | 31
days | 7.00 [6.00 to 14.00] | 7.00 [6.00 to 7.00]

10. Secondary Outcome: Area Under the Curve-During the Dosing Interval Tau (AUC [0-tau]) : Parallel-Arm Period
Description: AUC0-tau: area under the serum concentration versus time curve calculated using the trapezoidal method during a dosage interval tau, where dosing interval was 4 weeks.
Time Frame: Pre-dose (Week 0) and on Day 7, 14 and 21
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 32 | 31
ng*day/mL | 381000 (147000) | 414000 (152000)

11. Secondary Outcome: Maximum Serum Alirocumab Concentration Observed - Cmax : Single-Arm Period
Description: Cmax: maximum serum concentration observed.
Time Frame: Pre-dose (Week 4, Week 8 and Week 12) and on Day 7, 14, 21 and 28 days following the last injection
Population: Analysis was performed on PK population of the single-arm period which included all randomized participants who received at least 1 dose or part of a dose of IMP and had at least one evaluable blood sample for PK during this period. Here, "Overall number of participants analyzed" = participants evaluable for this PK measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | New Auto-injector Device (SYDNEY)
Number analyzed (Participants) | 64
ng/mL | 31900 (13100)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alirocumab: Single-Arm Period
Description: Tmax: Time to reach Cmax.
Time Frame: Pre-dose (Week 4, Week 8 and Week 12) and on Day 7, 14, 21 and 28 days following the last injection
Population: Analysis was performed on PK population of the single-arm period. Here, "Overall number of participants analyzed" = participants evaluable for this PK measure.
Measure: Median (Full Range); unit: days
Arm/Group | New Auto-injector Device (SYDNEY)
Number analyzed (Participants) | 64
days | 7.00 [3.00 to 11.00]

13. Secondary Outcome: Area Under the Curve-During the Dosing Interval Tau (AUC [0-tau]) : Single-Arm Period
Description: as for outcome 10
Time Frame: Pre-dose (Week 4, Week 8 and Week 12) and on Day 7, 14, 21 and 28 days following the last injection
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 63
ng*day/mL | 509000 (264000)

14. Secondary Outcome: Free Proprotein Convertase Subtilisin Kexin Type 9 (PCSK9) Concentrations : Parallel-Arm Period
Description: Free PCSK9 concentrations below the lower limit of quantification (LLOQ) were set to zero.
Time Frame: Week 4
Population: Analysis was performed on PK population of the parallel-arm period. Here, "Overall number of participants analyzed" = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 33 | 32
ng/mL | 90.1 (110.5) | 78.3 (103.1)

15. Secondary Outcome: Free Proprotein Convertase Subtilisin Kexin Type 9 (PCSK9) Concentrations : Single-Arm Period
Description: Free PCSK9 concentrations below the LLOQ were set to zero.
Time Frame: Week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 65
ng/mL | 88.9 (116.4)

16. Secondary Outcome: Total Proprotein Convertase Subtilisin Kexin Type 9 (PCSK9) Concentrations : Parallel-Arm Period
Description: Total PCSK9 concentrations below the LLOQ were set to zero.
Time Frame: Week 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 33 | 32
ng/mL | 3329.7 (1147.7) | 3370.0 (916.6)

17. Secondary Outcome: Total Proprotein Convertase Subtilisin Kexin Type 9 (PCSK9) Concentrations : Single-Arm Period
Description: Total PCSK9 concentrations below the LLOQ were set to zero.
Time Frame: Week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 65
ng/mL | 3481.4 (1290.1)

18. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Alirocumab Antibodies (ADA) Positive Response: Parallel-Arm Period
Description: Anti-drug (alirocumab) antibodies samples were analyzed using a validated electrochemiluminescence assay. Number of participants with positive ADA during treatment emergent adverse event (TEAE) period (time from the first IMP injection to the day before the second IMP injection for participants entered into the single arm period or to 70 days after the first IMP injection, whichever comes first) was determined. Treatment-emergent positive ADA response defined as 1) participants with no ADA positive response at baseline but with any positive response in the post-baseline period or 2) participants with a positive ADA response at baseline and at least a 4- fold increase in titer in the post-baseline period.
Time Frame: Up to Week 4
Population: Analysis was performed on ADA population of the parallel-arm period which included all randomized participants who received at least 1 or part of a dose of IMP during this period with baseline and at least one post-baseline available ADA sample during this period. All participants were analyzed according to the AI device they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 32 | 32
Participants | 2 | 1

19. Secondary Outcome: Number of Participants With Treatment-Emergent Anti-Alirocumab Antibodies (ADA) Positive Response According to ADA Status During Parallel-Arm Period: Single Arm Period
Description: Number of participants with positive ADA during the TEAE period (time from the second IMP injection up to the day of last IMP injection + 70 days) were determined. Treatment-emergent positive ADA response in Single-arm period defined as 1) participants with no ADA positive response in the Parallel-arm period but with any positive response in the Single-arm period or 2) participants with a positive ADA response at baseline, with less than 4-fold increase in titer in the Parallel-arm period (Pre-existing ADA in Parallel-arm period) and at least a 4- fold increase in titer in the Single-arm period.
Time Frame: Week 16
Population: Analysis was performed on ADA population of single-arm period which included all randomized participants who received at least 1 or partial dose of IMP during this period with available baseline and at least 1 post-baseline ADA sample available during this period. Here, "Number analyzed" = participants with ADA assessed at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 64
Participants
  Pre-existing ADA: number analyzed (Participants) | 1
  Pre-existing ADA | 0
  Negative ADA status: number analyzed (Participants) | 60
  Negative ADA status | 2
  Treatment-emergent ADA positive: number analyzed (Participants) | 3
  Treatment-emergent ADA positive | 0

20. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 4: Parallel-Arm Period
Description: Adjusted least square means and standard errors at Week 4 were calculated from analyses of covariance (ANCOVA) model with the fixed categorical effect of treatment group (SYDNEY, AI), as well as the continuous fixed covariate of baseline LDL-C value.
Time Frame: From Baseline to Week 4
Population: Analysis was performed on modified intent-to-treat (mITT) population of the parallel-arm period which included all randomized participants who received at least 1 dose or part of a dose of IMP during this period and who had an evaluable baseline and an on-treatment LDL-C value within Week 4 analysis window and before second injection, if any.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Auto-Injector Device (AI) | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 32 | 31
percent change | -51.2 (4.4) | -66.2 (4.4)

21. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 8, 12, 16: Single-Arm Period
Time Frame: From Baseline to Weeks 8, 12, and 16
Population: mITT population of single-arm period included all randomized participants who continued in single-arm period & received at least 1 dose/part of a dose of IMP & who had an evaluable baseline & at least 1 on-treatment LDL-C value within analysis windows (Week 8 to 16). Number analyzed=participants with available data at specified time-point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | New Auto-Injector Device (SYDNEY)
Number analyzed (Participants) | 66
percent change
  Week 8 | -53.737 (32.641)
  Week 12: number analyzed (Participants) | 65
  Week 12 | -58.610 (25.068)
  Week 16: number analyzed (Participants) | 64
  Week 16 | -56.991 (25.930)

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to final visit (Week 16) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment emergent that is AEs that developed/worsened during 'the treatment emergent period' (the time from first IMP injection to the second IMP injection for participants entering into the single-arm period, or to 70 days after first IMP injection, whichever comes first [Parallel arm period] or the time from the second IMP injection up to the day of last IMP injection + 70 days [Single arm period]). Analysis was performed on safety population.
Groups:
- Auto-Injector Device (AI) (Parallel Arm Period): Alirocumab 300 mg SC injection on Week 0 (Day 1), self-administered using AI device, on-site under supervision in the parallel arm period of 4 weeks added to LMT.
- New Auto-Injector Device (Parallel-arm Period): Alirocumab 300 mg SC injection on Week 0 (Day 1), self-administered using new auto-injector device (SYDNEY), on-site under supervision in the parallel arm period of 4 weeks added to LMT.
- New Auto-Injector Device (Single-arm Period): Alirocumab 300 mg SC injection on Week 0 (Day 1), self-administered using new auto-injector device (SYDNEY), on-site under supervision in the parallel arm treatment period of 4 weeks. From Week 4, same treatment (Alirocumab 300 mg) with the same device (SYDNEY) was self-administered, (unsupervised) Q4W at Week 4, 8 and 12 in the single arm treatment period. Duration of single arm treatment period was 12 weeks, i.e. from Week 4 to 16 added to LMT.
Arm/Group | Auto-Injector Device (AI) (Parallel Arm Period) | New Auto-Injector Device (Parallel-arm Period) | New Auto-Injector Device (Single-arm Period)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/33 | 2/66
Other Adverse Events (participants affected / at risk) | 2/34 | 5/33 | 8/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-Injector Device (AI) (Parallel Arm Period) (N=34) | New Auto-Injector Device (Parallel-arm Period) (N=33) | New Auto-Injector Device (Single-arm Period) (N=66)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Chondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-Injector Device (AI) (Parallel Arm Period) (N=34) | New Auto-Injector Device (Parallel-arm Period) (N=33) | New Auto-Injector Device (Single-arm Period) (N=66)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03415178/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT03415178/SAP_001.pdf